CLINICAL TRIAL: NCT06539468
Title: Investigating Active Surveillance for Management of Low-Risk Basal Cell Carcinoma in the Elderly
Brief Title: Active Surveillance for the Treatment of Low-Risk Basal Cell Carcinoma in Elderly Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2023.115; NCI-2024-05523 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HUM00243172 (Other: University of Michigan)
Record Dates: First submitted 2024-07-18; First posted 2024-08-06 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Skin Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Practice Guidelines as Topic; Standard of Care; Watchful Waiting; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part A (educational activity, survey administration) (Experimental): Patients watch an educational video on AS for LR-BCC and complete a survey about comfort with AS for LR-BCC on study.
  Interventions: Other: Educational Activity; Other: Survey Administration
- Part B arm 1 (active surveillance) (Active Comparator): Patients receive no treatment and undergo active surveillance over 1 year in the absence of disease progression. Patients may choose to undergo treatment at any point on study. Patients complete a standard 1-year follow-up total body skin examination followed by a second survey.
  Interventions: Other: Patient Observation; Other: Survey Administration
- Part B arm 2 (SOC) (Active Comparator): Patients receive SOC treatment which typically includes either electrodesiccation and curettage, surgical resection, or Mohs surgery as agreed upon by patient and provider in the absence of disease progression. Patients complete a standard 1-year follow-up total body skin examination followed by a second survey.
  Interventions: Other: Best Practice; Other: Survey Administration

INTERVENTIONS:
Other: Best Practice — Receive SOC treatment
  Other Names: standard of care; standard therapy
  Arms: Part B arm 2 (SOC)
Other: Educational Activity — Watch an educational video on AS for LR-BCC
  Arms: Part A (educational activity, survey administration)
Other: Patient Observation — Undergo active surveillance
  Other Names: Active Surveillance; deferred therapy; expectant management; Observation; Watchful Waiting
  Arms: Part B arm 1 (active surveillance)
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates whether active surveillance (AS) is a safe and comfortable alternative to standard of care (SOC) treatment for elderly patients with low-risk basal cell carcinoma (LR-BCC). Basal cell carcinoma is a type of slow-growing skin cancer that has a very low risk of spreading inside the body (metastasis) or death. Basal cell skin cancers that are smaller across than a nickel in size and located on the trunk or limbs are particularly low risk to overall health. Active surveillance - watching and not treating unless the cancer worsens - has been shown to be a generally safe way to manage LR-BCC. Despite this, many doctors do not feel comfortable discussing this option with patients due to a lack of studies comparing it to standard of care treatment. Standard of care treatment for LR-BCC can include "scrape and burn" (electrodesiccation and curettage), surgical resection, Mohs surgery, and other approaches. These treatments can carry risks like post-operative bleeding and wound infection, and they do not always improve tumor-related quality of life. Active surveillance may be a safe and comfortable alternative to SOC treatment for elderly patients with LR-BCC.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify the baseline characteristics of patients who are willing and able to enroll in an randomized controlled trial (RCT) examining acceptability of AS versus (vs.) SOC. (Part A) II. To determine if satisfaction of patients randomized to AS is noninferior to satisfaction of those randomized to SOC at one-year follow-up. (Part B)

EXPLORATORY OBJECTIVES:

I. To collect additional pilot data on acceptability of AS for asymptomatic LR-BCC among the elderly.

II. To determine the feasibility and optimal design of a future fully powered multi-institution RCT examining the hypothesis that active surveillance of biopsy-proven low-risk BCC is an acceptable alternative to standard treatment.

III. To collect pilot data on clinical outcomes of AS versus SOC for asymptomatic LR-BCC among the elderly for a duration of one year (the typical interval for skin cancer screening examinations for patients with a history of skin cancer).

IV. To compare the effects of AS vs. SOC for LR-BCC among the elderly on healthcare utilization.

V. To identify baseline characteristics that may predict a positive experience with AS.

VI. To explore perceived benefits of and concerns regarding participation in the RCT among the study population.

VII. To explore perceived benefits of and concerns regarding AS for LR-BCC among the study population.

VIII. To explore causes of nonadherence to maintenance of randomization in part B.

IX. To explore causes of nonadherence to follow-up in part B.

OUTLINE:

PART A: Patients watch an educational video on AS for LR-BCC and complete a survey about comfort with AS for LR-BCC on study.

PART B: Patients are randomized to 1 of 2 arms - as below and complete a standard 1-year follow-up total body skin examination followed by a second survey.

ARM 1: Patients receive no treatment and undergo active surveillance over 1 year in the absence of disease progression. Patients may choose to undergo treatment at any point on study.

ARM 2: Patients receive SOC treatment which typically includes either electrodesiccation and curettage, surgical resection, or Mohs surgery as agreed upon by patient and provider in the absence of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Subject of any gender aged ≥ 65 years at the time of enrollment
* Patient at University of Michigan Department of Dermatology (UMichDD)
* Willing and able to provide informed consent
* Willing and able to comply with the protocol requirements
* Histopathologic diagnosis of one or more LR-BCC(s) within 2 months of enrollment. LR-BCC is defined here as biopsy proven primary (not recurrent) BCC of any morphologic subtype; < 2cm in size; with or without marginal involvement on histopathology; and located on the trunk or extremities excluding pretibial surface, hands, feet, nail units, and ankles (corresponding to area L in the Mohs Appropriate Use Criteria, representing the lowest risk areas)

Exclusion Criteria:

* Individuals who are immunocompromised per judgement of investigator (examples include but are not limited to patients on immunosuppressive medications such as prednisone > 10 mg daily, uncontrolled HIV, and organ transplant recipients on immunosuppressive therapy)
* Individuals who expect to relocate and will be unable to return to UMichDD for clinical follow-up visit(s)
* Individuals with a genetic syndrome predisposing to development of basal cell carcinoma

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-12-28 (Estimated); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
Enrollment in part B (Part A) | 6 months
  Will evaluate the associations between baseline characteristics and the primary outcome of enrollment in part B (up to accrual target for 100 subjects) by logistic regression. Baseline characteristics include demographics, clinical data, patient-reported measures, baseline comfort with active surveillance (AS), and interest in enrollment in part B. The clinical research coordinator will assign each participant in part A a value of 1 if enrolled in part B or 0 if not enrolled (up to accrual target of 100 subjects for part B).
Satisfaction with AS/standard of care (SOC) (Part B) | At week 52
  Will compare the satisfaction of participants randomized to AS versus SOC as measured by five-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Billi, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States